CLINICAL TRIAL: NCT06945692
Title: Assessment of Accuracy and Aesthetics Following Automated Mandibular Defect Reconstruction Using Artificial Intelligence: A Case Series Study
Brief Title: Assessment of Accuracy and Aesthetics Following Automated Mandibular Defect Reconstruction Using AI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Moustafa Mahmoud Fahmy El-Youtti, Assistant lecturer, oral and maxillofacial surgery department, Ahram Canadian University, PHD Student at Cairo university., Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI in Mandibular Defects
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Mandibular Tumor
Keywords: Artificial intelligence; Patient specific reconstruction plates
MeSH Terms: conditions — Mandibular Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient specific reconstruction plates (Experimental): Patients with benign lesions indicated for resection and resulting in mandibular continuity defects treated with patient specific reconstruction plates.
  Interventions: Procedure: patient specific reconstruction plates

INTERVENTIONS:
Procedure: patient specific reconstruction plates — Use of patient specific reconstruction plates on the 3-D virtually-generated defect using Artificial Intelligence.

SUMMARY:
The Aim of the study is to evaluate Accuracy of automated mandibular defect reconstruction using Artificial intelligence and assessing impact on aesthetic and occlusion outcomes using patient-specific reconstruction plates.

DETAILED DESCRIPTION:
The digital surgical process often requires an expected mandibular reference model. Currently, the common digital surgery process, is to mirror repair or manually look for other similar mandibles for local data fusion and smoothing processing. A more accurate expected reference model is difficult to achieve, time consuming and difficult to promote in clinical practice. Moreover, rapid routing processing often has poor accuracy. For cumulative bilateral lesions, massive lesions, obvious displacement or lesions cross the middle line, there is still no effective method to predict the expected reference model in clinical practice.

The main objective for conducting this study is to propose an improved algorithm to overcome the drawbacks of recent studies using 3D Unet and to test the predictability and clinical value of virtually generated 3d models of defected mandible in real patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mandibular tumors, cysts or any benign disease resulting in mandibular continuity defect.
* Age group: from 18 - 55 years old.
* No sex predilection.
* CTs or CBCTs of only healthy mandibles from an online database and real data.

Exclusion Criteria:

* Patients with mandibular malignant lesions.
* Children age group from 2-17.
* CTs Of maxilla.
* Elderly patients to be excluded due to the normal physiologic bony change.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy Of the virtually Generated 3D model using AI | baseline
  The measuring device is the AI model using the Percentage as a unit
Accuracy of AI generated model clinically | baseline
  The measuring device is by Superimposition of both virtual 3-d generated model and real patient CT post operative using software ( blender ) .
  ( Structural Similarity Index) (SSIM)

SECONDARY OUTCOMES:
Aethetic outcome | baseline
  The measuring device is Facial appearance using a 4-point score
Occlusion | baseline
  The measuring device is Digital occlusion analysis using T-scan and the unit is percentage

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Moustafa, MSc., Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liang Y, Huan J, Li JD, Jiang C, Fang C, Liu Y. Use of artificial intelligence to recover mandibular morphology after disease. Sci Rep. 2020 Oct 2;10(1):16431. doi: 10.1038/s41598-020-73394-5. PMID 33009429
- [Background] van Baar GJC, Forouzanfar T, Liberton NPTJ, Winters HAH, Leusink FKJ. Accuracy of computer-assisted surgery in mandibular reconstruction: A systematic review. Oral Oncol. 2018 Sep;84:52-60. doi: 10.1016/j.oraloncology.2018.07.004. Epub 2018 Jul 20. PMID 30115476